CLINICAL TRIAL: NCT00832338
Title: Phase II Trial of Pre-Operative Docetaxel-Cytoxan (TC) in Patients With Hormone Receptor-Positive Cancers With Recurrence Scores ≥ 25
Brief Title: Trial Using Docetaxel Cytoxan in Breast Cancers With High Recurrence Scores
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding withdrawn
Sponsor: Emory University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Elisavet Paplomata, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00012185; WCI1505-08 (Other: Other)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Breast Neoplasms; Breast Cancer; Cancer of the Breast
Keywords: Breast cancer; Tumors, Breast; Cancer of the breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Cyclophosphamide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel with Cytoxan (Experimental): Patients will be treated with docetaxel at 75 mg/m² concomitantly with cytoxan 600 mg/m² (TC) IV D1 every 3 weeks for 6 cycles. Due to known toxicity of docetaxel, all patients require dexamethasone 4 mg twice daily (BID) PO for 3 consecutive days starting 12-24 hours prior to each dose of docetaxel to minimize hypersensitivity reactions and fluid retention.
  Interventions: Drug: Docetaxel with Cytoxan; Drug: Dexamethasone

INTERVENTIONS:
Drug: Docetaxel with Cytoxan — Docetaxel 75 mg/m² plus cytoxan 600 mg/m² every 3 weeks for 6 cycles.
  Other Names: Docetaxel; Cytoxan
Drug: Dexamethasone — Dexamethasone 4 mg BID PO for 3 consecutive days starting 12-24 hours prior to each dose of docetaxel.
  Other Names: Decadron

SUMMARY:
The purpose of this study is to assess if docetaxel and cytoxan can shrink the size of your breast tumor and allow you to preserve your breast or have less extensive surgery on your breast. Additionally, by receiving chemotherapy before surgery, the investigators will be able to determine if your cancer is responsive to chemotherapy.

DETAILED DESCRIPTION:
Previous studies have shown that chemotherapy has the same effect on treating breast cancer whether you receive it before or after surgery. Receiving chemotherapy before surgery, rather than after surgery, may allow you to have less extensive surgery by shrinking the size of your cancer. The purpose of this study is to assess if docetaxel and cytoxan can shrink the size of your breast tumor and allow you to preserve your breast or have less extensive surgery on your breast. Additionally, by receiving chemotherapy before surgery, we will be able to determine if your cancer is responsive to chemotherapy. Prior to entering this study, a special test, called the Oncotype DX assay, will be performed on a small amount of your cancer from the biopsy you had at the time you were diagnosed with breast cancer, to determine the likelihood that your cancer will benefit from and shrink with chemotherapy. You will only be eligible to enter this study if the recurrence score determined using the Oncotype DX assay is 25 or greater. Patients with hormone receptor-positive breast cancers with recurrence scores greater than or equal to 25 have been previously demonstrated to obtain a significant benefit from chemotherapy given after surgery.

In addition, researchers would like to examine proteins present in your blood and proteins present in your breast tissue. These additional parts of the study are voluntary and are NOT required to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Histologically or cytologically confirmed breast carcinoma.
* Early stage breast cancer (T1c-3, clinically node-negative-3 [cN0-3], cM0).
* No evidence of disease outside the breast or chest wall, except ipsilateral axillary or internal mammary lymph nodes.
* Pre-treatment biopsy with the following characteristics:

  * Hormone receptor-positive cancer as defined as ER and/or progesterone receptor (PR)-positive by standard immunohistochemistry (IHC)
  * HER2-negative (HER2 ≤ 2 by IHC; if HER2 2+ by IHC must be fluorescence in situ hybridization [FISH] non-amplified)
  * Recurrence score ≥ 25 using Oncotype DX 21-gene assay
* Patients must have measurable disease as defined by palpable lesion with both diameters ≥ 1cm measurable with caliper or a positive mammogram or ultrasound with at least one dimension ≥ 1cm. Baseline measurements of the indicator lesions must be recorded on the Patient Registration Form. To be valid for baseline, the measurements must have been made within the 14 days if palpable. If not palpable, a mammogram or MRI must be done within 14 days. If palpable, a mammogram or MRI must be done within 2 months prior to study entry. If clinically indicated, xrays and scans must be done within 28 days of study entry.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2.
* No prior chemotherapy, hormonal therapy, biologic therapy or radiation therapy for breast cancer.
* Adequate organ function within 14 days of study entry:

  * Bone marrow function: absolute neutrophil count (ANC) ≥ 1500/mm³, Hgb > 8.0 g/dl, and platelet count ≥ 100,000/mm³.
  * Hepatic function: total bilirubin < upper limit of normal (ULN). Serum glutamic oxaloacetic transaminase (SGOT)(AST) or serum glutamic pyruvic transaminase (SGPT)(ALT) and alkaline phosphatase ≤ 1.5 x ULN.
  * Renal function: calculated creatinine clearance (CrCl) ≥ 30 mL/min using the Cockroft Gault equation.
* Patients must be at least 18 years of age.

Exclusion Criteria:

* Pregnant or lactating women are not eligible. Women of childbearing potential must have a negative serum pregnancy test completed within 7 days of study entry, and use an appropriate form of birth control throughout the trial period.
* No medical, psychological or surgical condition which the investigator feels might compromise study participation.
* No patients with history within the last 5 years of previous or current malignancy at other sites with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies who remain disease free for greater than five years are eligible.
* No evidence of peripheral or sensory neuropathy.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 are excluded from participation.
* No serious, uncontrolled, concurrent infection(s).
* No clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months prior to study entry.
* No major surgery within 28 days of study entry.
* No evidence of central nervous system (CNS) metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisavet Paplomata, MD, Principal Investigator — Emory University Winship Cancer Institute
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Winship Cancer Institute, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from April 2009 to October 2015 at Winship Cancer Institute of Emory University, Emory University Hospital Midtown, and Grady Memorial Hospital.
Period: Overall Study
Arm/Group | Docetaxel With Cytoxan
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Docetaxel With Cytoxan: Patients will be treated with docetaxel at 75 mg/m² concomitantly with cytoxan 600 mg/m² (TC) IV D1 every 3 weeks for 6 cycles. Due to known toxicity of docetaxel, all patients require dexamethasone 4 mg BID PO for 3 consecutive days starting 12-24 hours prior to each dose of docetaxel to minimize hypersensitivity reactions and fluid retention.
  Docetaxel with Cytoxan: Docetaxel 75 mg/m² plus cytoxan 600 mg/m² every 3 weeks for 6 cycles.
  Dexamethasone: Dexamethasone 4 mg BID PO for 3 consecutive days starting 12-24 hours prior to each dose of docetaxel.
Arm/Group | Docetaxel With Cytoxan
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.91 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 20
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response to Pre-operative Docetaxel and Cytoxan (TC)
Description: Patients were assessed for surgery after 6 cycles of TC (18 weeks). Pathologic stage was determined based on size of tumor and degree of lymph node involvement at the time of surgery, whereas clinical stage pre-operatively was determined by clinical assessment and imaging.
  If pathologic stage was the same as clinical stage, it was called stable; if it was higher, upstaged (worse outcome); if lower, downstaged (better outcome). Pathologic stage was determined by Emory board-certified pathologists.
Time Frame: At time of definitive surgery
Population: Staging information was not collected for two patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Docetaxel With Cytoxan
Number analyzed (Participants) | 21
Participants
  Downstaged | 12
  Stable | 4
  Upstaged | 5

ADVERSE EVENTS:
Arm/Group | Docetaxel With Cytoxan
Serious Adverse Events (participants affected / at risk) | 1/23
Other Adverse Events (participants affected / at risk) | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel With Cytoxan (N=23)
Febrile neutropenia (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Docetaxel With Cytoxan (N=23)
Dyspepsia (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Syncope (Nervous system disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Increased creatinine (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Pruritis (Skin and subcutaneous tissue disorders) | 1
Irregular menstruation (Reproductive system and breast disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Weight gain (General disorders) | 2
Fatigue (General disorders) | 16
Tachycardia (Cardiac disorders) | 1
Nail loss (Skin and subcutaneous tissue disorders) | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 6
Myalgias (Musculoskeletal and connective tissue disorders) | 2
Maculopapular rash (Skin and subcutaneous tissue disorders) | 5
Watery eyes (Eye disorders) | 3
Upper respiratory infection (Infections and infestations) | 1
Abdominal pain (General disorders) | 1
Memory impairment (Nervous system disorders) | 1
Anorexia (Gastrointestinal disorders) | 3
Sensory peripheral neuropathy (Nervous system disorders) | 12
Alopecia (Skin and subcutaneous tissue disorders) | 8
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 4
Lower extremity edema (Blood and lymphatic system disorders) | 8
Oral mucositis (Gastrointestinal disorders) | 4
Dysgeusia (Gastrointestinal disorders) | 6
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8
Insomnia (General disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Anxiety (Psychiatric disorders) | 5
Depression (Psychiatric disorders) | 3
Mood swings (Psychiatric disorders) | 1
Allergic reaction (Immune system disorders) | 1
Headache (Nervous system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes